CLINICAL TRIAL: NCT06858878
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Maridebart Cafraglutide in Adult Participants With Type 2 Diabetes Mellitus Who Have Obesity or Are Overweight (MARITIME-2)
Brief Title: Efficacy and Safety of Maridebart Cafraglutide in Adult Participants With Type 2 Diabetes Mellitus Who Have Obesity or Are Overweight
Acronym: MARITIME-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210184
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM), Obesity, Overweight
Keywords: Type 2 Diabetes Mellitus; T2DM; Obesity; Overweight; Maridebart Cafraglutide; AMG 133; MariTide; Chronic Weight Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Maridebart Cafraglutide High Dose (Experimental): Participants will receive maridebart cafraglutide high dose subcutaneously (SC) for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Maridebart Cafraglutide Medium Dose (Experimental): Participants will receive maridebart cafraglutide medium dose SC for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Maridebart Cafraglutide Low Dose (Experimental): Participants will receive maridebart cafraglutide low dose SC for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Maridebart cafraglutide will be adminstered SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide High Dose; Maridebart Cafraglutide Low Dose; Maridebart Cafraglutide Medium Dose
Drug: Placebo — Placebo will be adminstered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate that maridebart cafraglutide is superior to placebo for percent change in body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Body mass index ≥ 27 kg/m^2.
* History of at least 1 self-reported unsuccessful attempt at weight loss by diet and exercise.
* Diagnosis of T2DM.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Self-reported change in body weight > 5 kg within 90 days before screening.
* Proliferative diabetic retinopathy OR diabetic macular edema OR non-proliferative diabetic retinopathy that requires acute treatment.
* Obesity induced by other endocrinologic disorders.
* Family (first-degree relative[s]) or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2.
* History of chronic pancreatitis or history of acute pancreatitis within 180 days before screening.
* History of unstable major depressive disorder (MDD) or other severe psychiatric disorder within 2 years before screening.
* Lifetime history of suicide attempt.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight at Week 72 | Baseline and Week 72

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference at Week 72 | Baseline and Week 72
Participant achieving ≥ 5% reduction in body weight from baseline at week 72 | Baseline and Week 72
Participant achieving ≥ 10% reduction in body weight from baseline at week 72 | Baseline and Week 72
Participant achieving ≥ 15% reduction in body weight from baseline at week 72 | Baseline and Week 72
Change from Baseline in Systolic Blood Pressure (SBP) at Week 72 | Baseline and Week 72
Percent Change from Baseline in Fasting Triglycerides at Week 72 | Baseline and Week 72
Change from Baseline in Fasting Plasma Glucose at Week 72 | Baseline and Week 72
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 72 | Baseline and Week 72
Participant achieving HbA1c < 7% at week 72 | Week 72
Change from Baseline in the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score at Week 72 | Baseline and Week 72
Change from Baseline in Body Weight at Week 72 | Baseline and Week 72
Participant achieving ≥ 20% reduction in body weight from baseline at week 72 | Baseline and Week 72
Change from Baseline in Body Mass Index (BMI) at Week 72 | Baseline and Week 72
Participant achieving HbA1c ≤ 6.5% at week 72 | Week 72
Participant achieving HbA1c < 5.7%, at week 72 | Week 72
Percent Change from Baseline in Fasting Insulin at Week 72 | Baseline and Week 72
Percent Change from Baseline in High-sensitivity C-reactive Protein (hs-CRP) at Week 72 | Baseline and Week 72
Change from Baseline in Urine Albumin-to-creatinine Ratio (uACR) at Week 72 | Baseline and Week 72
Percent Change from Baseline at Week 72 in Fasting Concentration of Total Cholesterol | Baseline and Week 72
Percent Change from Baseline at Week 72 in Fasting Concentration of Non-high-density Lipoprotein Cholesterol (non-HDL-C) | Baseline and Week 72
Percent Change from Baseline at Week 72 in Fasting Concentration of Low-density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 72
Percent Change from Baseline at Week 72 in Fasting Concentration of Very-low-density Lipoprotein Cholesterol (VLDL-C) | Baseline and Week 72
Percent Change from Baseline at Week 72 in Fasting Concentration of High-density Lipoprotein Cholesterol (HDL-C) | Baseline and Week 72
Change from Baseline in Diastolic Blood Pressure DBP at Week 72 | Baseline and Week 72
Change from Baseline in Short Form 36 Health Survey Version 2 (SF-36v2) Acute Physical Function Domain Score at Week 72 | Baseline and Week 72
Number of Participants who Experienced Treatment-emergent Adverse Events | Up to Week 84
Number of Participants who Experienced Serious Adverse Events | Up to Week 84
Plasma Concentration of Maridebart Cafraglutide at Week 72 | Week 72

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (186):
- United States (58):
  - Alliance for Multispecialty Research Mobile, Mobile, Alabama
  - Gilbert Center for Family Medicine, Gilbert, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Avacare Foothills Research Center, Phoenix, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - Core Healthcare Group, Cerritos, California
  - Velocity Clinical Research Chula Vista, Chula Vista, California
  - Headlands Research California, Escondido, California
  - Paradigm Clinical Research, Modesto, California
  - Flourish Research, Northridge, California
  - University of California Irvine, Orange, California
  - Empire Clinical Research, Pomona, California
  - Infinity Clinical Trials, San Diego, California
  - Greenwich Clinical Trials, Riverside, Connecticut
  - Indago Research and Health Center, Hialeah, Florida
  - Optimus U Corporation, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Encore Medical Research of Weston LLC, Weston, Florida
  - Conquest Research - Winter Park, Winter Park, Florida
  - Alliance For Multispecialty Research - Oak Brook, Oak Brook, Illinois
  - Alliance for Multispecialty Research, LLC - Park Ridge, Park Ridge, Illinois
  - Endeavor Health Medical Group - Endocrinology and Diabetes- Skokie, Skokie, Illinois
  - Indiana Medical Research Institute, Merrillville, Indiana
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Alliance for Multispecialty Research Newton, Newton, Kansas
  - Alliance for Multispecialty Research LLC, Wichita, Kansas
  - Advanced Internal Medicine, Paducah, Kentucky
  - Ima Clinical Research- Monroe, Monroe, Louisiana
  - Annapolis Internal Medicine, LLC, Annapolis, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - International Diabetes Center - HealthPartners Institute, Minneapolis, Minnesota
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Palm Research Center Inc, Las Vegas, Nevada
  - Vector Clinical Trials, Sparks, Nevada
  - Premier Research, Trenton, New Jersey
  - Albany Medical College, Albany, New York
  - Asheville Clinical Research, Asheville, North Carolina
  - Physicians East, Greenville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Velocity Clinical Research - Cincinnati, Blue Ash, Ohio
  - Velocity Clinical Research - Springdale, Cincinnati, Ohio
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Medical Care LLC, Elizabethton, Tennessee
  - Elligo Clinical Research Center, Austin, Texas
  - Osvaldo A Brusco MD PA, Corpus Christi, Texas
  - Cedar Health Research, LLC, Dallas, Texas
  - Soma Clinical Trials, LLC, Denison, Texas
  - Cedar Health Research, LLC, Euless, Texas
  - Juno Research LLC, Houston, Texas
  - Tekton Research, McKinney, Texas
  - Northeast Clinical Research of San Antonio LLC, San Antonio, Texas
  - Alliance for Multispecialty Research - Layton, Layton, Utah
  - Manassas Clinical Research Center Inc, Manassas, Virginia
  - VA Puget Sound Healthcare System, Seattle, Washington
  - Ima Clinical Research - West Virginia, Morgantown, West Virginia
- Argentina (7):
  - Centro Medico Viamonte, CABA, Buenos Aires
  - Cedic Centro de Investigacion Clinica, CABA, Buenos Aires
  - Cemedic Centro de Especialidades Medicas, CABA, Buenos Aires
  - Maffei Centro Medico, CABA, Buenos Aires
  - Consultorios Medicos Dr Besada, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Ciprec Centro de Investigacion y Prevencion Cardiovascular, Ciudad Autonoma de Buenos Aires, Buenos Aires
- Bulgaria (6):
  - Ambulatory for specialized outpatient medical aid in endocrinology-Dr Albena Dinkova EOOD, Pleven
  - Diagnostic - Consultative Center XX - Sofia EOOD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed OOD, Sofia
  - Prevencia-2000-Medical center for outpatient medical aid OOD, Stara Zagora
  - Medical Center Berbatov EOOD, Yambol
- Canada (19):
  - tlc Diabetes and Endocrinology, Surrey, British Columbia
  - Chronic Disease Innovation Centre, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Queen Elizabeth ii Health Sciences Centre, Halifax, Nova Scotia
  - Centricity Research Brampton, Brampton, Ontario
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Centricity Research Vaughan, Concord, Ontario
  - Winterberry Family Medicine, Hamilton, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Centricity Research Ottawa LMC, Nepean, Ontario
  - Your Research Network Inc., Niagara Falls, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Bluewater Clinical Research Group Incorporated, Sarnia, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Centricity Research Quebec City, Lévis, Quebec
  - Institut de recherches cliniques de Montreal, Montreal, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Centricity Research Pointe-Claire, Pointe-Claire, Quebec
  - Diex Recherche Trois Rivieres, Trois-Rivières, Quebec
- Czechia (11):
  - Fakultni nemocnice Brno, Brno
  - CCR Ostrava sro, Ostrava
  - Diahelp sro, Pardubice
  - Pratia Pardubice as, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Milan Kvapil sro, Prague
  - Restrial sro, Prague
  - Endokrinologie Cerny Most sro, Prague
  - Milan Kvapil sro, Pribram VIII
- Germany (20):
  - Universitatsklinikum Aachen, Aachen
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Diabetespraxis Bad Mergentheim, Bad Mergentheim
  - Universitaetsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Velocity Clinical Research GmbH, Berlin
  - Diabetespraxis Dr. Hermann Braun, Berlin
  - Mvz am Bahnhof Spandau, Berlin
  - Zentrum fuer Klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung, Essen
  - Schwerpunktpraxis fuer Diabetes, Gefaess- & Ernaehrungsmedizin, Falkensee
  - Diabeteszentrum Hamburg West, Hamburg
  - Endokrinologikum Hamburg, Hamburg
  - Diabetologische Schwerpunktpraxis Hohenmoelsen, Hohenmölsen
  - Universitaetsklinikum Leipzig, Leipzig
  - AmBeNet GmbH, Leipzig
  - Kardiologische Praxis Doktor Jens Taggeselle, Markkleeberg
  - Centrum für Diagnostik und Gesundheit, München
  - Zentrum fuer Diabtes und Gefaesskrankheiten im Franziskus Carré Muenster, Münster
  - Red-Institut GmbH, Oldenburg
- Hungary (11):
  - Lausmed Kft, Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - ClinDiab Kft, Budapest
  - MED-TIMA Kft, Budapest
  - Borvo Clinic Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Komaromi Selye Janos Korhaz, Komárom
  - Borbanya Praxis Egeszsegugyi Kft, Nyíregyháza
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Italy (7):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Sacco, Milan
  - Ospedale Civico, Di Cristina e Benfratelli, Palermo
- Japan (11):
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama, Ehime
  - Morizono Medical Clinic, Kitakyusyu-shi, Fukuoka
  - Mazda Hospital of Mazda Motor Corporation, Aki-gun, Hiroshima
  - Nakamoto Medical Clinic, Mito, Ibaraki
  - Nakakinen Clinic, Naka, Ibaraki
  - Ohishi Naika Clinic, Tsuchiura-shi, Ibaraki
  - Morinaga Ueno Clinic, Kumamoto, Kumamoto
  - Shiraiwa Medical Clinic, Kashiwara-shi, Osaka
  - Suruga Clinic, Shizuoka, Shizuoka
  - Yutenji Medical Clinic, Meguro-ku, Tokyo
  - Medical Corporation Ouitsukai Kanno Naika, Mitaka-shi, Tokyo
- Poland (12):
  - Salvia-Lekston i Madej Spolka Jawna, Katowice
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa Gabinet Lekarski, Lublin
  - Ekamed Spolka z Ograniczona Odpowiedzialnoscia, Lublin
  - Medicome Spolka z Ograniczona Odpowiedzialnoscia, Oświęcim
  - Velocity Nova Sp zoo Velocity Pulawy, Puławy
  - NZOZ Przychodnia Specjalistyczna A Wittek H Rudzki spolka jawna, Ruda Śląska
  - Velocity Nova Sp zoo Velocity Staszow, Staszów
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - Nbr Polska Tomasz Klodawski, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Wromedica I Bielicka A Strzalkowska SC, Wroclaw
- Latin Clinical Trial Center, San Juan, Puerto Rico
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - KyungHee University Gangdong Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- United Kingdom (11):
  - Ormeau Clinical Trials Ltd, Belfast
  - FutureMeds Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - Waterloo Medical Centre, Blackpool
  - Southmead Hospital, Bristol
  - Staploe Medical Centre, Ely
  - FutureMeds Glasgow, Glasgow
  - Hull Royal Infirmary, Hull
  - NIHR Leicestershire & Northamptonshire Commercial Research Delivery Centre, Leicester
  - Aintree University Hospital, Liverpool
  - Clifton Medical Centre, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com